CLINICAL TRIAL: NCT03282734
Title: Effect of the Home-based Exercise Program With Smart Rehabilitation System on Balance and Gait Functions in Stroke Patients
Brief Title: Home-based Exercise Program With Smart Rehabilitation System
Acronym: Smart-Rehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-07-072
Record Dates: First submitted 2017-09-10; First posted 2017-09-14 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The smart rehab group (Experimental): Home-based exercise program with smart rehabilitation system ((Uincare®, D-gate Co.) for 4 weeks
  Interventions: Other: Home-based exercise program with smart rehabilitation system ((Uincare®, D-gate Co.)
- The control group (Active Comparator): Conventional home rehabilitation exercise education for 4 weeks
  Interventions: Other: Conventional home rehabilitation exercise

INTERVENTIONS:
Other: Home-based exercise program with smart rehabilitation system ((Uincare®, D-gate Co.) — Home-based exercise program with smart rehabilitation system ((Uincare®, D-gate Co.) for more than 30 minutes per a day for 4 weeks
  Arms: The smart rehab group
Other: Conventional home rehabilitation exercise — Conventional home rehabilitation exercise for more than 30 minutes per a day for 4 weeks
  Arms: The control group

SUMMARY:
A lot of patients suffer the balance and gait disorders after stroke. Many rehabilitation therapies have been provided to improve the balance and gait function in stroke patients. However, most rehabilitation therapies are performed in only hospitals, in spite of the difficulty of moving from home to hospitals for stroke patients. Home-based smart rehabilitation system (Uincare®, D-gate Co.) can provide the specific rehabilitation training program to stroke patients in their home. This study aims to investigate the effects of the home-based exercise program with smart rehabilitation system on balance and gait functions in stroke patients.

DETAILED DESCRIPTION:
The total 100 patients with stroke will be divided into each the intervention group and the control group. The intervention group will be provided the home-based smart rehabilitation system for 4 weeks, and the control group will be educated the conventional home rehabilitation exercise at once. The immediate effects of the home-based smart rehabilitation system on the balance and gait function will be assessed at 4 weeks after exercise and the long-term carry-over effects will be also assesed at 4 weeks after cessation of exercise.

ELIGIBILITY:
Inclusion Criteria:

* adult stroke patients (more than 18 years old)
* less than 6 months after stroke onset
* discharged to home or the plan to discharge to home less than 3 days
* independent ambulatory function on even level (4 or more than 4 in Functional Ambulatory Category)

Exclusion Criteria:

* Advanced liver, kidney, cardiac, or pulmonary disease
* A terminal medical diagnosis consistent with survival < 1 year)
* Pre-existing and active major neurological disease
* Pre-existing and active major psychiatric disease
* Severe language disorders
* Severe cognitive disorders (10 or less than 10 in K-MMSE)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go test | Change from baseline Timed Up and Go test at 4 weeks
  Assessment of balance and gait function

SECONDARY OUTCOMES:
Tinetti Performance Oriented Mobility Assessment | Change from baseline Timed Up and Go test at 4 weeks
  Assessment of balance and gait function
Berg Balance scale | Change from baseline Timed Up and Go test at 4 weeks
  Assessment of balance
Korean-Geriatric Depression Scale- Short Form | Change from baseline Timed Up and Go test at 4 weeks
  Assessment of mood
EQ-5D | Change from baseline Timed Up and Go test at 4 weeks
  Assessment of quality of life
Falls Efficacy Scale | Change from baseline Timed Up and Go test at 4 weeks
  Assessment of fall risk
Korean version of Physical Activity Scale for the Elderly | Change from baseline Timed Up and Go test at 4 weeks
  Assessment of physical activity

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No